CLINICAL TRIAL: NCT03764657
Title: Pilonidal Sinus Disease: Preliminary Case-control Study on Heat-related Wound Dehiscence
Brief Title: Pilonidal Sinus Disease: Preliminare Study
Status: Completed | Type: Observational
Sponsor: Ospedale di Cavalese (Other)
Responsible Party: Sponsor
Other Study IDs: OCavalese172018
Record Dates: First submitted 2018-11-25; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Pilonidal Sinus
Keywords: Pilonidal sinus disease; wound deiscence
MeSH Terms: conditions — Pilonidal Sinus | interventions — Cold Temperature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 16 patients, named "Hot" group: We considered 16 sinus excision by diathermy as a case group (named "Hot" group)
  Interventions: Procedure: In "hot" group 16 patients were treated by diathermy in "Cold"; Procedure: in "Cold" group 13 patients were treated by scalpel.
- 13 patients, named "Cold group": 13 procedures performed by knife as control group (named "Cold" group).
  Interventions: Procedure: In "hot" group 16 patients were treated by diathermy in "Cold"; Procedure: in "Cold" group 13 patients were treated by scalpel.

INTERVENTIONS:
Procedure: In "hot" group 16 patients were treated by diathermy in "Cold" — In all interventions, the patients were placed in prone position on operating table with the gluteal line opened wide by adhesive patches; after skin disinfection, dimension and extension of cystic disease was studied by injection of hydrogen peroxide through superficial skin orifice. The same procedure was performed: an elliptical incision on midline around the sinus was made and the sinus was excided laterally and in depth on healthy tissue, down till the pre-sacral fascia: this common approach was made both using scalpel and electrosurgery in the two groups. During dissection and excision, in each group were measured and recorded the temperatures developing, both on the section surface using an infrared thermometer and thermal imaging camera, and deeper until 1 cm from the section frontline using a "immersion thermometer" sealed by a steri-drape to guarantee the sterility on surgical field. In this group excision was carried out with diatermocoagulation
Procedure: in "Cold" group 13 patients were treated by scalpel. — the position and preparation of the patient on the operating table were the same as in the "hot" group, while the excision procedure performed with knife

SUMMARY:
Pilonidal disease is morbid condition of young productive population, that could impair quality of life with high cost for health care system. No consensus exists on optimal surgical treatment, even if several techniques have been proposed. In this preliminary experimental case-control study the investigators compared excision by knife and diathermy with the aim to investigate if wound dehiscence could be related to heat spreading during excision of the sinus.

DETAILED DESCRIPTION:
Between January 2017 and February 2018, 29 patients underwent to sinus excision. The investigators considered 16 sinus excision performed by diathermy as a case group (named "Hot" group) and the last 13 procedures performed by knife as control group (named "Cold" group). Temperature data were recorded for both group. Follow-up was carried out until complete healing. Were considered primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients between 14 and 65 years old,
* primary, non recurrent pilonidal disease
* midline and intergluteal location
* spinal anesthesia
* dimension no more than 5 cm in length, primary closure performed

Exclusion Criteria:

* age < 14 and > 65 years old,
* secondary fistulous tracts or lateral developing/cutaneous opening
* dimension over 5 cm in length,
* local anesthesia employ
* smoker and obese patients (BMI> 25 kg/m2)
* diabetic and coagulopathies affected one
* flogged or acute or infected or abscessed forms
* ASA score > IV,
* normal range WBC and Hb preoperative values.

Ages: 14 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients were enrolled by outpatient surgical control for signs and symptoms of chronic sinus referred to us by a family doctor; median age was 19.2 ± 4.3 years, ranging from 14 to 52 years old; 6 patients were females and 23 males and them were request to give informed consensus to underwent to pilonidal sinus excision; 16 patients of whom 12 males and 4 females, were treated by electrosurgery as case group ("hot"), while in the control group ("cold"), 13 patients 11 were male and 2 were females.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of complete wound healed and not healed after 8 postoperative days | Up to 4 weeks
  We established as primary outcomes, the number of wound completely healed after 8-12 days

SECONDARY OUTCOMES:
types of complications (Dindo-Clavien) | follow-up 12 months
  the type of complication was divided into 2 types, Grade I and II
post-operative pain in first postoperative day (analogue pain score, VAS) | 7 days
  postoperative pain was recorded in the two groups using the analog pain scale (VAS, range 0-10, the lowest value indicates less pain and the highest value indicates)
operative time for complete excision of the sinus (minutes) | minutes (range 0-30 minutes)
  the operative time for complete excision was compared into the two group

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale di Cavalese, Cavalese, Trento, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Giuseppe F, Silvia DG, Patrizia R, Riccardo P, Antonio DS, Aldo RS, Angela I, Pietro M, Domenico M, Luciano T. Pilonidal sinus disease: Preliminary case-control study on heat-related wound dehiscence. Ann Med Surg (Lond). 2019 Aug 18;48:144-149. doi: 10.1016/j.amsu.2019.07.032. eCollection 2019 Dec. PMID 31890195